CLINICAL TRIAL: NCT05291325
Title: Application of Linaclotide Capsule in Bowel Preparation for Colonoscopy: a Multicenter, Randomized, Controlled Clinical Study
Brief Title: Application of Linaclotide Capsule in Bowel Preparation for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Shanxi Provincial People's Hospital (Other Government); 900 Hospital of Joint Logistics Support Force of PLA (Other); Ruijin Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); Qilu Hospital of Shandong University (Other); The Affiliated Hospital of Qingdao University (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); Affiliated Yueqing Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Soochow University (Other); The 7th Medical Center of the PLA General Hospital (Unknown); The First Hospital of Jilin University (Other); The Second Hospital of Hebei Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Ningxia Medical University General Hospital (Unknown); Affiliated Hospital of Qinghai University (Other); Yunnan First People's Hospital (Unknown); Second Xiangya Hospital of Central South University (Other); Shanghai Zhongshan Hospital (Other); Daping Hospital, Army Military Medical University (Unknown); Zunyi Medical College (Other); Huizhou Municipal Central Hospital (Other); Affiliated Hospital of Southwest Medical University (Other); The First Hospital of Shihezi University (Unknown); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tangdu Hospital of Air Force Military Medical University (Unknown)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Linaclotide
Record Dates: First submitted 2022-03-18; First posted 2022-03-22 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Bowel Preparation for Colonoscopy
Keywords: Linaclotide; Bowel preparation; colonoscopy
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3L PEG + Linaclotide (Experimental): Bowel preparation for colonoscopy was performed with 3L polyethylene glycol solution combined with 3-day linaclotide.
  Interventions: Drug: 3L PEG + Linaclotide
- 3L PEG alone (Active Comparator): Bowel preparation for colonoscopy was performed with 3L polyethylene glycol solution without linaclotide.
  Interventions: Drug: 3L PEG
- 2L PEG + Linaclotide (Experimental): Bowel preparation for colonoscopy was performed with 2L polyethylene glycol solution combined with 3-day linaclotide.
  Interventions: Drug: 2L PEG + Linaclotide

INTERVENTIONS:
Drug: 3L PEG + Linaclotide — Before colonoscopy, particpant take linaclotide capsules for 3 days (1 tablet should be taken at least 30 minutes before the first meal every day). Particpant take 1500ml polyethylene glycol electrolyte solution within 1.5 hours from 20 p.m the night before the examination; and repeat the same dose of polyethylene glycol electrolyte solution 4-6 hours before colonoscopy.
  Arms: 3L PEG + Linaclotide
Drug: 3L PEG — Particpant take 1500ml polyethylene glycol electrolyte solution within 1.5 hours from 20 p.m the night before the examination; and repeat the same dose of polyethylene glycol electrolyte solution 4-6 hours before colonoscopy.
  Arms: 3L PEG alone
Drug: 2L PEG + Linaclotide — Before colonoscopy, particpant take linaclotide capsules for 3 days (1 tablet should be taken at least 30 minutes before the first meal every day). Particpant take 1000ml polyethylene glycol electrolyte solution within 1 hours from 20 p.m the night before the examination; and repeat the same dose of polyethylene glycol electrolyte solution 4-6 hours before colonoscopy.
  Arms: 2L PEG + Linaclotide

SUMMARY:
The clinical purpose of this study was to investigate whether the adjuvant application of linaclotide in bowel preparation for colonoscopy could improve the quality of bowel preparation or reduce the dosage of laxatives.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, male or female;
* To undergo diagnostic, screening or monitoring colonoscopy;
* Signed written informed consent;

Exclusion Criteria:

* Severe cardiopulmonary insufficiency, renal failure or a history of stroke or myocardial infarction within six months;
* History of abdominal or pelvic surgery;
* Pregnant and lactating women;
* BMI > 28, BMI < 18.5, inflammatory bowel disease, constipation (defecation less than 3 times in the last week, and laborious defecation, fecal sclerosis, low volume) or intestinal obstruction and other high-risk factors of intestinal preparation;
* Abnormal coagulation function or taking antiplatelet or anticoagulant drugs within 7 days;
* Warning symptoms and signs of colorectal cancer: hematochezia, melena, unexplained anemia, low body weight, abdominal mass, positive digital rectal test; or imaging and laboratory tests highly suspect colorectal cancer;
* Colon polyps have been identified;
* Stow score 7 (watery, no solid mass), diarrhea was considered;
* Participation in other interventional clinical trials within 60 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1607 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Bowel preparation adequate rate | within 10 minute after viewing colonoscopy video.
  The proportion of participants with all colon segment scores (right colon, transverse colon, left colon) were ≥ 2 according to Boston Bowel Preparation Scale (BBPS) .

SECONDARY OUTCOMES:
Boston bowel preparation scale score | Within 10 minute after viewing colonoscopy video.
  The BBPS scoring rules: 0, unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared; 1, portion of mucosa of the colon segment seen, but other areas of the colon segment are not well seen because of staining, residual stool, and/or opaque liquid; 2, minor amount of residual staining, small fragments of stool, and/or opaque liquid, but mucosa of colon segment is seen well; 3, entire mucosa of colon segment seen well, with no residual staining, small fragments of stool, or opaque liquid. the higher the score, the better the quality of bowel preparation. 3 intestinal segments were scored separately: the right side of the colon, the transverse section of the colon, and the left side of the colon. Total BBPS score 0-9, the higher the score, the better the quality of bowel preparation.
Aronchick Scale | Within 10 minute after viewing colonoscopy video.
  Overall bowel preparation was scored prior to irrigation or suction. The Aronchick Scale scoring rules: 1, excellent, a small amount of liquid, 95% mucous membrane is visible; 2, good, plenty of clear fluid, covering 5%-25% of mucous membrane, 90% mucous membrane is visible; 3, medium, semi-solid manure that cannot be sucked out or washed away, 90% mucous membrane is visible; 4, poor, semi-solid manure that cannot be sucked out or washed away, 90% mucous membrane is visible; 5, inadequate, repeated bowel preparation or reexamination is required. Total Aronchick score 1-5, the lower the score, the better the quality of bowel preparation.
Bowel preparation excellent rate | Within 10 minute after viewing colonoscopy video.
  The proportion of participants with total score ≥ 8 according to Boston Bowel Preparation Scale.
Bowel preparation completion rate assessed by questionnaire survey | Immediately after questionnaire survey.
  Proportion of subjects with laxative intake greater than 90% of the required amount in protocol.
Subjects satisfaction rate assessed by questionnaire survey | Immediately after questionnaire survey.
  Proportion of subjects satisfacted with the whole intestinal preparation process. Subjects satisfaction was divided into four grades: 4, very satisfied; 3, moderately satisfied; 2, moderately dissatisfied; 1, very dissatisfied. Subjects in grades 3 and 4 were considered satisfied; subjects in grades 1 and 2 were considered dissatisfied.
Endoscopists satisfaction with the quality of bowel preparation | Immediately after colonoscopy.
  Proportion of endoscopists satisfacted with the quality of bowel preparation during colonoscopy. Endoscopists satisfaction was divided into four grades: 4, very satisfied; 3, moderately satisfied; 2, moderately dissatisfied; 1, very dissatisfied. Subjects in grades 3 and 4 were considered satisfied; subjects in grades 1 and 2 were considered dissatisfied.
Adenoma detection rate | 14 days after colonosopy.
  The adenoma detection rate was calculated as the number of colonoscopies with at least one adenoma detected divided by the total number of colonoscopies in the group. Adenomatous polyps must be confirmed by pathological findings.
Polyp detection rate | Immediately after colonoscopy.
  The polyp detection rate was calculated as the number of colonoscopies with at least one polyp detected divided by the total number of colonoscopies in the group.
Incidence of adverse events assessed by questionnaire survey | Immediately after questionnaire survey.
  Proportion of subjects with adverse events occuring in intestinal preparation.
Drug compliance in linaclotide group | Immediately after questionnaire survey.
  Proportion of subjects Taking 3 linaclotide capsules according to the protocol in linaclotide group.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Naval Medical University, Shanghai, China

REFERENCES:
- [Background] Zhang M, Zou W, Xu C, Jia R, Liu K, Xu Q, Xu H. Polyethylene glycol combined with linaclotide is an effective and well-tolerated bowel preparation regimen for colonoscopy: an endoscopist-blinded, randomized, controlled trial. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e625-e633. doi: 10.1097/MEG.0000000000002184. PMID 34034273
- [Derived] Pan P, Chen H, Wang T, Liu K, Tuo B, Wang R, Fu H, Jiang C, Chen L, Zhao Q, Wang W, Chen W, Guo Q, Chen W, Li Y, Tian Z, Feng Z, Yang S, Fan Y, Luan F, Chen Y, Li Z, Bai Y. Effect of 3-Day Linaclotide Administration to Reduce the Polyethylene Glycol Volume for Colonoscopy Bowel Preparation: A Multicenter, Noninferiority, Randomized Controlled Trial. Am J Gastroenterol. 2025 May 27. doi: 10.14309/ajg.0000000000003557. Online ahead of print. PMID 40423516